CLINICAL TRIAL: NCT01253226
Title: Multiple-Dose, Dose-Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LY2127399 in Japanese Patients With Rheumatoid Arthritis Treated With Methotrexate
Brief Title: A Study for Japanese Participants With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13060; H9B-JE-BCDK (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tabalumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 30 milligrams (mg) Tabalumab (Experimental): 30 mg tabalumab every 4 weeks (Q4W) for 20 weeks (6 doses of study drug)
  Interventions: Drug: LY2127399 (Tabalumab)
- 60 mg Tabalumab (Experimental): 60 mg tabalumab Q4W for 20 weeks (6 doses of study drug)
  Interventions: Drug: LY2127399 (Tabalumab)
- 120 mg Tabalumab (Experimental): 120 mg tabalumab Q4W for 20 weeks (6 doses of study drug)
  Interventions: Drug: LY2127399 (Tabalumab)
- Placebo Q4W (Placebo Comparator): Q4W for 20 weeks
  Interventions: Drug: Placebo
- 120 mg once every 2 weeks (Q2W) Tabalumab (Experimental): Initial loading dose of 240 mg tabalumab followed by 120 mg Q2W for 20 weeks (10 doses of study drug)
  Interventions: Drug: LY2127399 (Tabalumab)
- Placebo Q2W (Placebo Comparator): Q2W for 20 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2127399 (Tabalumab) — Administered subcutaneously
  Other Names: LY2127399; Tabalumab
  Arms: 120 mg Tabalumab; 120 mg once every 2 weeks (Q2W) Tabalumab; 30 milligrams (mg) Tabalumab; 60 mg Tabalumab
Drug: Placebo — Administered subcutaneously
  Arms: Placebo Q2W; Placebo Q4W

SUMMARY:
This study will evaluate the safety and tolerability of multiple doses of LY2127399 (tabalumab) in Japanese participants with RA. The study consists of a 20-week treatment period. All participants will be followed for up to 12 weeks after the last study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Women must not be pregnant, breastfeeding or be at risk to become pregnant during study participation
* Diagnosis of RA
* Active RA
* Current, regular use of Methotrexate, at a stable dose
* Body weight between 40 and 105 kilograms (kg), inclusive

Exclusion Criteria:

* Use of excluded medications (reviewed by study doctor)
* Have medical findings which, in the opinion of the study doctor, put participant at an unacceptable risk for participation in the study
* Have had recent or ongoing infection which, in the opinion of the study doctor put participant at an unacceptable risk for participation
* Evidence of tuberculosis
* Have systemic inflammatory condition other than RA

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM-5 PM Eastern time (UTC/GMT - 5 hours, EST ), Study Director — Eli Lilly and Company
Locations (10):
- Japan (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukui
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This dose-escalation study had 4 cohorts. Each cohort included 6 LY2127399 (tabalumab) participants and 2 placebo participants. Participants treated once every 2 weeks (Q2W) or once every 4 weeks (Q4W) and had a follow-up visit at Week 32. Additional visits beyond Week 32 were scheduled, as needed, for B cell count monitoring (up to 12 weeks).
Groups:
- 30 mg Tabalumab Q4W: Tabalumab: 30 milligrams (mg) subcutaneous (SC) injection Q4W for 20 weeks (Weeks 0, 4, 8, 12, 16, and 20).
- 60 mg Tabalumab Q4W: Tabalumab: 60 mg SC injection Q4W for 20 weeks (Weeks 0, 4, 8, 12, 16, and 20).
- 120 mg Tabalumab Q4W: Tabalumab: 120 mg SC injection Q4W for 20 weeks (Weeks 0, 4, 8, 12, 16, and 20).
- 120 mg Tabalumab Q2W: Tabalumab: 240 mg SC injection given as a loading dose at Week 0 followed by 120 mg SC injection Q2W for 20 weeks (Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, and 20).
- Placebo: Q4W cohorts: Placebo SC injection Q4W for 20 weeks (Weeks 0, 4, 8, 12, 16, and 20).
  Q2W cohort: Placebo SC injection Q2W for 20 weeks (Weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, and 20).
Period: Overall Study
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W | Placebo
Started | 6 | 6 | 6 | 6 | 8
Received at Least 1 Dose of Study Drug | 6 | 6 | 6 | 6 | 8
Completed | 6 | 5 | 5 | 5 | 6
Not Completed | 0 | 1 | 1 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least 1 dose of study drug (tabalumab or placebo).
Groups:
- 30 mg Tabalumab Q4W: Tabalumab: 30 mg SC injection Q4W for 20 weeks (Weeks 0, 4, 8, 12, 16, and 20).
- Total: Total of all reporting groups
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (5.9) | 50.0 (15.0) | 55.5 (14.2) | 56.7 (8.0) | 58.4 (17.1) | 57.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 4 | 7 | 25
  Male | 0 | 2 | 2 | 2 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 6 | 6 | 6 | 6 | 8 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 6 | 6 | 6 | 6 | 8 | 32
Current Use of Corticosteroids [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 1 | 4 | 6 | 15
  No | 3 | 5 | 5 | 2 | 2 | 17
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 54.8 (5.5) | 55.9 (13.8) | 55.9 (10.5) | 58.3 (8.3) | 54.6 (7.5) | 55.8 (8.9)
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — CRP is an indicator of inflammation. Higher values indicate a greater amount of inflammation
  milligrams per deciliter (mg/dL) | 11.46 (13.90) | 18.69 (35.23) | 14.91 (9.17) | 8.73 (8.26) | 11.07 (5.30) | 12.85 (16.56)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) [Clinically Significant Effects]
Description: Clinically significant effects are defined as serious AEs (SAEs) and other non-serious AEs regardless of causality. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through study completion (up to Week 32 plus up to 12 weeks for B cell monitoring)
Population: Randomized participants who received at least 1 dose of study drug (tabalumab or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants
  SAEs, all causes | 0 | 1 | 1 | 1 | 1
  Non-Serious AEs, all causes | 5 | 4 | 3 | 6 | 5

2. Secondary Outcome: Pharmacokinetics (PK) of Tabalumab: Area Under the Concentration Time Curve (AUC)
Description: The following parameters are reported for the first SC injection of tabalumab: AUC(0-tlast) defined as AUC from time 0 to time t, where t is the time at the end of the dosing interval; AUC(0-2W) defined as AUC from time 0 to Week 2; and AUC(0-tau) defined as AUC during 1 dosing interval at steady state.
Time Frame: Week 0: Day 1 [predose and 1 hour (h), 3 h, and 6 h postdose], Days 2, 3, and 5, and Weeks 1, 2, 3, and 4 postdose
Population: Randomized participants who received at least 1 dose of tabalumab and had evaluable AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day/milliliter (mcg*day/mL)
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W
Number analyzed (Participants) | 6 | 6 | 6 | 6
micrograms*day/milliliter (mcg*day/mL)
  AUC(0-tlast) | 57.0 (24) | 148 (38) | 303 (49) | 303 (30)
  AUC(0-2W): number analyzed (Participants) | 6 | 6 | 6 | 5
  AUC(0-2W) | 30.3 (26) | 86.5 (34) | 170 (46) | 280 (35)
  AUC(0-tau): number analyzed (Participants) | 5 | 1 | 4 | 5
  AUC(0-tau) | 55.5 (27) | 173 (NA) — Only 1 participant included in the analysis, therefore the geometric coefficient of variation is not calculable. | 260 (58) | 280 (35)

3. Secondary Outcome: PK of Tabalumab: Maximum Observed Drug Concentration (Cmax)
Description: Cmax for the first SC injection of tabalumab is reported.
Time Frame: Week 0: Day 1 Predose, 1 h, 3 h, and 6 h postdose
Population: Randomized participants who received at least 1 dose of tabalumab and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W
Number analyzed (Participants) | 6 | 6 | 6 | 6
micrograms per milliliter (mcg/mL) | 2.88 (26) | 7.61 (35) | 16.6 (61) | 25.0 (28)

4. Secondary Outcome: Percent Change From Baseline in B Cell [Cluster Designation 20+ (CD20+)] Counts
Description: B-lymphocyte antigen, CD20+, is an activated-glycosylated phosphoprotein expressed on the surface of all mature B cells. Percent change from baseline in B cell counts=[(post-baseline CD20+ B cell count-baseline CD20+ B cell count)/(baseline CD20+ B cell count)]*100. A negative change indicates a decrease in cell count.
Time Frame: Baseline, Week 0 (Day 2), Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, and 32
Population: Randomized participants who received at least 1 dose of study drug (tabalumab or placebo) and had a baseline and at least 1 post-baseline B cell assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 7
percent change
  Week 0 (Day 2) | 13.7 (20.7) | 15.6 (60.0) | 16.1 (22.5) | 13.7 (34.4) | 34.9 (49.9)
  Week 1: number analyzed (Participants) | 6 | 6 | 6 | 5 | 5
  Week 1 | 42.8 (25.8) | 82.1 (107.8) | 100.7 (91.2) | 55.3 (53.9) | -7.2 (8.7)
  Week 2: number analyzed (Participants) | 6 | 6 | 6 | 4 | 6
  Week 2 | 14.9 (34.5) | 48.2 (80.2) | 73.0 (58.8) | 53.7 (12.9) | -12.0 (41.4)
  Week 3: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
  Week 3 | 7.7 (33.7) | 45.4 (63.3) | 65.7 (63.5) | 43.1 (23.3) | 0.3 (38.7)
  Week 4: number analyzed (Participants) | 6 | 6 | 6 | 5 | 5
  Week 4 | -12.1 (36.7) | 31.0 (81.6) | 46.1 (58.4) | 13.1 (32.1) | 5.5 (22.2)
  Week 6: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
  Week 6 | 6.7 (42.8) | 10.9 (65.9) | 67.7 (69.4) | 48.9 (43.2) | 2.1 (44.6)
  Week 8: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
  Week 8 | -10.3 (37.3) | 2.2 (57.0) | 36.7 (58.6) | 5.9 (46.0) | 2.9 (32.2)
  Week 12: number analyzed (Participants) | 6 | 6 | 6 | 4 | 6
  Week 12 | -17.6 (31.7) | -0.4 (76.3) | 22.8 (60.7) | 10.0 (38.6) | -7.0 (24.7)
  Week 16: number analyzed (Participants) | 6 | 6 | 5 | 4 | 6
  Week 16 | -24.7 (32.4) | -37.9 (27.1) | 27.0 (74.1) | -8.3 (29.2) | 0.6 (35.2)
  Week 20: number analyzed (Participants) | 6 | 6 | 5 | 4 | 6
  Week 20 | -30.4 (32.8) | -17.1 (59.1) | 54.1 (72.6) | -13.4 (30.7) | 2.5 (65.1)
  Week 24: number analyzed (Participants) | 6 | 5 | 3 | 4 | 6
  Week 24 | -34.4 (32.3) | -51.7 (25.9) | 26.4 (76.3) | -30.4 (26.3) | -2.9 (44.4)
  Week 32: number analyzed (Participants) | 6 | 5 | 5 | 4 | 4
  Week 32 | -59.0 (17.9) | -50.7 (36.1) | -17.9 (31.1) | -38.7 (17.8) | -4.0 (37.0)

5. Secondary Outcome: Change From Baseline in Anti-Cyclic Citrullinated Peptide (Anti-CCP) Antibody [Inova Enzyme-Linked Immunosorbent Assay (ELISA) Method]
Description: During the analysis of anti-CCP, the analytical method was changed from the Inova ELISA method to the Roche Cobas 6000 method due to the discontinuation of a reagent used in the Inova ELISA method. The anti-CCP data are summarized separately for samples collected before and after the method change. No post-baseline samples from the 120 mg tabalumab Q4W and Q2W cohorts were analyzed using the Inova ELISA method. For both methods, a decrease in anti-CCP antibodies indicated an improvement in the participant's condition.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of study drug (tabalumab or placebo) and had a baseline and at least 1 post-baseline anti-CCP assessment using the Inova ELISA method. No participants were analyzed in the 120 mg tabalumab Q4W and Q2W cohorts.
Measure: Mean (Standard Deviation); unit: units (U)
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W | Placebo
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 3
units (U) | -63.3 (138.8) | 63.3 (337.0) |  |  | 9.3 (58.2)

6. Secondary Outcome: Change From Baseline in Anti-CCP Antibody (Roche Cobas 6000 Method)
Description: During the analysis of anti-CCP, the analytical method was changed from the Inova ELISA method to the Roche Cobas 6000 method due to the discontinuation of a reagent used in the Inova ELISA method. The anti-CCP data are summarized separately for samples collected before and after the method change. No baseline samples from the 30 mg, 60 mg, and 120 mg tabalumab Q4W cohorts were analyzed using the Roche Cobas 6000 method. For both methods, a decrease in anti-CCP antibodies indicated an improvement in the participant's condition.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of study drug (tabalumab or placebo) and had a baseline and at least 1 post-baseline anti-CCP assessment using the Roche Cobas 6000 method. No participants were analyzed in the 30 mg, 60 mg, and 120 mg tabalumab Q4W cohorts.
Measure: Median (Full Range); unit: units per milliliter (U/mL)
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 1
units per milliliter (U/mL) |  |  |  | NA [0.0 to 35.5] — Only 2 participants included in the analysis, therefore median is not calculable. | NA [0.0 to 0.00] — Only 1 participant included in the analysis, therefore median is not calculable.

7. Secondary Outcome: Change From Baseline in Rheumatoid Factor (RF)
Description: RF is an autoantibody (antibody directed against an organism's own tissues) most relevant in rheumatoid arthritis (RA). Higher RF levels indicate an aggressive RA and a higher risk of joint damage. A decrease in RF levels indicate an improvement in the participant's condition.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of study drug (tabalumab or placebo) and had a baseline and at least 1 post-baseline RF level assessment.
Measure: Mean (Standard Deviation); unit: kilo units per liter (kU/L)
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 7
kilo units per liter (kU/L) | -38.6 (23.2) | 29.6 (143.9) | -108.0 (97.0) | -41.5 (45.0) | -12.9 (76.2)

8. Secondary Outcome: Change From Baseline in Serum Immunoglobulins (IgG, IgM, IgA)
Description: Immunoglobulins, or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Change from baseline serum immunoglobulin G (IgG), immunoglobulin M (IgM), and immunoglobulin A (IgA) levels are reported. A negative change indicates a decrease in immunoglobulin levels.
Time Frame: Baseline, Weeks 4, 16, 24, and 32
Population: Randomized participants who received at least 1 dose of study drug (tabalumab or placebo) and had a baseline and at least 1 post-baseline serum immunoglobulin assessment.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
grams per liter (g/L)
  IgG, Week 4 | -0.1 (1.6) | 0.0 (0.7) | 0.5 (2.5) | -0.6 (1.0) | -0.1 (1.0)
  IgG, Week 16: number analyzed (Participants) | 6 | 6 | 5 | 5 | 7
  IgG, Week 16 | -2.2 (1.0) | -0.2 (2.6) | -1.4 (1.0) | -1.8 (1.4) | -0.3 (1.5)
  IgG, Week 24: number analyzed (Participants) | 6 | 6 | 5 | 5 | 7
  IgG, Week 24 | -2.4 (1.1) | -0.7 (2.8) | -2.1 (2.5) | -0.8 (0.8) | -0.1 (1.9)
  IgG, Week 32: number analyzed (Participants) | 6 | 5 | 5 | 5 | 6
  IgG, Week 32 | -2.1 (1.3) | -0.9 (2.4) | -2.7 (2.1) | -0.9 (1.2) | 0.4 (3.0)
  IgM, Week 4 | -0.2 (0.5) | -0.1 (0.1) | -0.2 (0.1) | -0.1 (0.0) | -0.1 (0.2)
  IgM, Week 16: number analyzed (Participants) | 6 | 6 | 5 | 5 | 7
  IgM, Week 16 | -0.4 (0.6) | -0.3 (0.3) | -0.2 (0.2) | -0.2 (0.1) | -0.1 (0.1)
  IgM, Week 24: number analyzed (Participants) | 6 | 6 | 5 | 5 | 7
  IgM, Week 24 | -0.6 (0.7) | -0.3 (0.2) | -0.3 (0.3) | -0.2 (0.1) | -0.1 (0.1)
  IgM, Week 32: number analyzed (Participants) | 6 | 5 | 5 | 5 | 6
  IgM, Week 32 | -0.6 (0.8) | -0.3 (0.3) | -0.4 (0.1) | -0.2 (0.1) | -0.1 (0.1)
  IgA, Week 4 | -0.1 (0.2) | -0.2 (0.2) | -0.4 (0.3) | -0.1 (0.4) | -0.3 (0.4)
  IgA, Week 16: number analyzed (Participants) | 6 | 6 | 5 | 5 | 7
  IgA, Week 16 | -0.6 (0.3) | -0.4 (0.2) | -0.5 (0.2) | -0.3 (0.4) | -0.3 (0.3)
  IgA, Week 24: number analyzed (Participants) | 6 | 6 | 5 | 5 | 7
  IgA, Week 24 | -0.7 (0.2) | -0.5 (0.3) | -0.6 (0.4) | -0.4 (0.3) | -0.3 (0.4)
  IgA, Week 32: number analyzed (Participants) | 6 | 5 | 5 | 5 | 6
  IgA, Week 32 | -0.7 (0.4) | -0.5 (0.4) | -0.7 (0.4) | -0.3 (0.2) | -0.3 (0.4)

9. Secondary Outcome: Percent Change From Baseline in CRP
Description: CRP is an indicator of inflammation. The percent change from baseline in CRP=[(post-baseline CRP- baseline CRP)/(baseline CRP)]*100. A negative change indicates an improvement in the participant's condition.
Time Frame: Baseline, Weeks 4, 8, 16, and 24
Population: Randomized participants who received at least 1 dose of study drug (tabalumab or placebo) and had a baseline and at least 1 post-baseline CRP assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 7
percent change
  Week 4 | 210.8 (624.0) | -16.0 (53.1) | -8.5 (56.7) | 16.8 (111.9) | 42.9 (85.0)
  Week 8 | -54.0 (16.6) | 18.1 (126.4) | 167.0 (537.9) | 31.6 (85.9) | -13.8 (59.5)
  Week 16: number analyzed (Participants) | 6 | 6 | 5 | 5 | 7
  Week 16 | -38.1 (76.3) | 840.8 (2138.7) | -83.1 (15.0) | -41.3 (15.4) | 19.8 (120.8)
  Week 24: number analyzed (Participants) | 6 | 6 | 5 | 5 | 7
  Week 24 | -55.9 (43.9) | -33.5 (40.8) | -75.5 (36.4) | 119.9 (147.7) | 39.6 (89.3)

10. Secondary Outcome: Percent Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Reference ranges are gender-specific and can vary slightly among laboratories. The normal range is approximately ≤10 millimeters per hour (mm/h) for males and ≤20 mm/h for females. Higher scores indicate greater inflammation. The percent change from baseline in ESR=[(post-baseline ESR- baseline ESR)/(baseline ESR)]*100. A decrease in ESR indicates an improvement in the participant's condition.
Time Frame: Baseline, Weeks 4, 8, 16, and 24
Population: Randomized participants who received at least 1 dose of study drug (tabalumab or placebo) and had a baseline and at least 1 post-baseline ESR assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
percent change
  Week 4 | -5.9 (31.8) | -22.0 (22.4) | -7.5 (32.4) | 11.7 (28.4) | 6.1 (30.8)
  Week 8 | -27.5 (22.1) | -23.3 (24.7) | -3.1 (55.9) | 8.9 (33.3) | 13.3 (49.4)
  Week 16: number analyzed (Participants) | 6 | 6 | 5 | 5 | 7
  Week 16 | -26.1 (38.2) | -28.7 (25.0) | -47.4 (27.4) | -18.4 (16.4) | -3.0 (41.6)
  Week 24: number analyzed (Participants) | 6 | 6 | 5 | 5 | 7
  Week 24 | -40.7 (20.4) | -42.4 (26.4) | -56.4 (28.1) | 22.3 (64.2) | 26.3 (56.7)

ADVERSE EVENTS:
Time Frame: Baseline through study completion (up to Week 32 plus up to 12 weeks for B cell monitoring)
Arm/Group | 30 mg Tabalumab Q4W | 60 mg Tabalumab Q4W | 120 mg Tabalumab Q4W | 120 mg Tabalumab Q2W | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 1/6 | 1/6 | 1/8
Other Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 3/6 | 6/6 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 mg Tabalumab Q4W (N=6) | 60 mg Tabalumab Q4W (N=6) | 120 mg Tabalumab Q4W (N=6) | 120 mg Tabalumab Q2W (N=6) | Placebo (N=8)
EYE MOVEMENT DISORDER (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OCULAR HYPERTENSION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STRABISMUS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA LEGIONELLA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONJUNCTIVAL ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 30 mg Tabalumab Q4W (N=6) | 60 mg Tabalumab Q4W (N=6) | 120 mg Tabalumab Q4W (N=6) | 120 mg Tabalumab Q2W (N=6) | Placebo (N=8)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GOITRE (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHALAZION (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
PERIODONTITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INJECTION SITE ERYTHEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (3)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD URINE PRESENT (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 0/4 (0) | 0/4 (0) | 1/4 (1) | 0/7 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1/4 (1) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHEUMATOID VASCULITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The anti-CCP data were difficult to interpret and compare for trends due to the 2 different methods of analysis used and the high variability in the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days